CLINICAL TRIAL: NCT01390025
Title: Phase 1 Study of TCN-032 (Human Monoclonal Antibody Directed Against the M2 Protein of Influenza A Virus) in Healthy Adult Volunteers
Brief Title: Safety Study of Anti-Influenza Virus Monoclonal Antibody to Treat Influenza
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theraclone Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TCN-032-001
Record Dates: First submitted 2011-07-05; First posted 2011-07-08 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2012-03

CONDITIONS: Influenza, Human
Keywords: Influenza; Monoclonal antibody
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TCN-032 (Experimental)
  Interventions: Biological: TCN-032
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: TCN-032 — TCN-032 is a human monoclonal antibody that specifically binds to a conserved epitope of the amino-terminal extracellular domain (M2e) of the influenza virus matrix protein 2 (M2). The drug is intended for use as an antiviral agent for the treatment of disease caused by type A influenza viruses. Treatments within the study will consist of single ascending dose-escalation ranging from 1 to 40 mg/kg.
  Arms: TCN-032
Biological: Placebo — Placebo - 0.9% Sodium Chloride for Injection, USP
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the safety profile in healthy volunteers of a single intravenous administration of TCN-032 as compared with placebo.

DETAILED DESCRIPTION:
Influenza is a highly communicable acute respiratory disease that is considered to be one of the major infectious disease threats to the human population. Annual vaccination is generally effective only against those strains included in the vaccine. Because of the frequent emergence of divergent variants and the periodic emergence of strains with novel hemagglutinin and/or neuraminidase surface proteins that can result in global pandemics, the availability of potent antiviral agents for the prevention and/or treatment of influenza remains an urgent clinical and public health priority.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Normal lab tests

Exclusion Criteria:

* Prior treatment with a monoclonal antibody

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Safety assessment - number of participants with adverse events (AE) | 60 days post infusion
  Safety will be assessed by physical examinations, vital signs, serial electrocardiograms and clinical laboratory tests (hematology, chemistry and urinalysis). A clinically significant laboratory value will be any abnormal result that is an unexpected or unexplained laboratory value or change in value from the patient's prior values. AEs will be reported by severity and relatedness to study treatment and classified according to MedDRA

SECONDARY OUTCOMES:
Pharmacokinetic analysis (PK)- Evaluate the single, ascending dose PK of TCN-032 | 60 days post infusion
  PK evaluation of TCN-032 plasma concentrations will include: tmax (time at which maximum concentration is observed),Cmax (maximum observed concentration), t1/2 (terminal-elimination half-life), CL (clearance), Vd (volume of distribution).
Immunogenicity - detect and measure generation of anti-drug antibodies (ADA)specific for TCN-032 | 60 days post infusion
  Immunogenicity will be assessed based on induction of TCN-032 anti-drug antibodies. Baseline and serial post-treatment serum measures of anti-TCN-032 antibodies will be detected by immunoassay and summarized by dose and time point with means, standard deviations, medians, quartiles, and ranges. Change from baseline in anti-TCN-032 antibody levels will be similarly analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Al-Ibrahim, MD, FACP, Principal Investigator — SNBL
Locations (1):
- SNBL Clinical Pharmacology Center, Baltimore, Maryland, United States

REFERENCES:
- [Background] Grandea AG 3rd, Olsen OA, Cox TC, Renshaw M, Hammond PW, Chan-Hui PY, Mitcham JL, Cieplak W, Stewart SM, Grantham ML, Pekosz A, Kiso M, Shinya K, Hatta M, Kawaoka Y, Moyle M. Human antibodies reveal a protective epitope that is highly conserved among human and nonhuman influenza A viruses. Proc Natl Acad Sci U S A. 2010 Jul 13;107(28):12658-63. doi: 10.1073/pnas.0911806107. Epub 2010 Jul 1. PMID 20615945